CLINICAL TRIAL: NCT06345053
Title: Presence of PTSD and Emotion Dysregulation Among Inpatients With Substance Use Disorder; a Feasibility Study of a Combined Treatment for Difficulties in Emotion Regulation and PTSD
Brief Title: Presence of PTSD and Emotion Dysregulation Among Inpatients With Substance Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Møre og Romsdal Hospital Trust (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 203428
Record Dates: First submitted 2024-03-06; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Post Traumatic Stress Disorder; Substance Use Disorders; Emotion Regulation; Suicide; Self-harm
Keywords: Dialectical Behaviour Therapy; Narrative Exposure Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Emotional Regulation; Suicide; Self-Injurious Behavior | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Intervention Model Description: This is a repeated measures follow-up feasibility study without control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trauma fit inclusion / accept participation in DBT-SUD skills NET (Experimental): All patients with relevant will be offered to participate in DBT-SUD skills training and or NET.
  Interventions: Behavioral: Narrative Exposure Therapy

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — The intervention period will be from (May 2021- October 2024). All patients will participate in standard treatment at MBS. Dialectical Behaviour Therapy -Substance Use Disorder skills training (DBT-SUD skills) will be offered to all patients at MBS in the project period that experience difficulties in emotion regulation and manage to commit to participating in the DBT- skills training evaluated by their DBT therapist. Narrative Exposure Therapy (NET) will be offered to all patients with relevant traumatic experience and symptoms of PTSD depending on clinical evaluation.
  Other Names: Dialectical Behaviour Therapy

SUMMARY:
There are high rates of co-occurring posttraumatic stress disorder (PTSD) among patients receiving treatment for substance use disorder (SUD). PTSD and SUD should be treated simultaneously, but adults in SUD treatment are often not assessed for PTSD nor offered PTSD-based interventions. One of the reasons for reluctance in offering trauma focused treatment is increased risk of drop out. PTSD and related emotion dysregulation are related to elevated psychological burden, higher dropout rates and increased risk of relapse. this is a feasibility study, where the plan is to integrate a combination of Dialectical Behaviour Therapy for Substance Use Disorder (DBT-SUD skills) a therapy targeting difficulties in emotion regulation and Narrative Exposure Therapy (NET) a trauma focused therapy, for patients with co-occurring PTSD symptoms into standard SUD treatment . The plan is to assess its potential benefits by assessing whether adding this combination to standard SUD treatment is relevant, feasible, acceptable, and safe. Treatment outcomes are 1) Prevalence of PTSD, suicidal behaviour, and self-harm, as well as the severity of difficulties in emotion regulation and emotional avoidance among patients (N approx. = 100) in inpatient treatment for SUD. 2) Change post-treatment and at 3 and 12 months follow up, from baseline in PTSD symptom severity, depressive symptoms, emotion regulation, emotion avoidance, and experience of shame. 3) Rates of dropout and relapse compared to previous rates.

This project can increase knowledge about psychological mechanisms in co-occurring PTSD and SUD and improve the quality of treatment for this vulnerable patient population.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria for the study:

  1. Fit general inclusion criteria for the in-patient program.
  2. Speak Scandinavian (Norwegian, Danish and/or Swedish).
  3. Be willing to sign a consent.

Inclusion criteria for NET intervention:

1. Experience of an aversive event that fits criteria A for PTSD as defined by Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V) (American Psychiatric Association [APA], 2013).
2. Experience symptoms of PTSD as defined by the DSM-V (APA, 2013), or subthreshold PTSD (Grubaugh et al., 2005), or experience clinically relevant symptoms as evaluated by a NET therapist.

   1. Subthreshold PTSD is defined as having experienced a traumatic event (Criteria A), meeting Criteria B (re-experiencing symptoms), Criteria E (one-month symptom duration), and Criteria F (significant distress or functioning impairment) and either Criteria C (avoidance or numbing symptoms) or Criteria D (hyper arousal symptoms).

Inclusion criteria for DBT intervention:

1. Experience difficulties in emotion regulation evaluated by an assigned DBT therapist.
2. Manage to commit to participating in the DBT- skills training.

Exclusion Criteria:

* General exclusion criteria for the study:

  1. Have a clinically significant low cognitive- and/or linguistic functioning that hinders the patient in understanding and answering the questions on the self-rapport instruments.

Exclusion criteria for NET and/or DBT-SUD skills

1. Being actively psychotic.
2. Have a Body Mass Index (BMI) under 17.
3. Severe dissociation.
4. An ongoing traumatic contact with the perpetrator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
The intervention is relevant - prevalence of PTSD /SUP PTSD. | One time assessment 5 weeks after admission to treatment
  The prevalence of PTSD/SUB-PTSD is measured with the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) a 30-item structured interview used to make current (past month) diagnosis of PTSD, make lifetime diagnosis of PTSD, and assess PTSD symptoms over the past week (Weathers et al., 2018). Frequency and intensity rating is summed to create an overall PTSD symptom severity score and is used to generate a categorical diagnosis (PTSD/Sub-PTSD vs non-PTSD). In this project, we will both use the categorical diagnosis to compare those with and without PTSD/Sub-PTSD, as using the overall PTSD symptom severity scores (Weathers et al., 2018).
The intervention is relevant - prevalence of traumatic experiences. | One time assessment 5 weeks after admission to treatment
  The prevalence of traumatic experiences also as offenders is measured with Stressful Life Events Screening Questionnaire-Revised (SLESQ) is self-report instrument designed to map and assess 15 potentially traumatic experiences (Goodman et al., 1998). The score is used to identify experiences of potential traumatic events. For this project, items asking about experiences where the participant caused potentially traumatic experiences to others are added. This is to identify violent offenders.
The intervention is relevant - The severitiy of difficulties in emotion regulation. | One time assessment 5 weeks after admission to treatment
  The severity of difficulties in emotion regulation will be measured with Difficulties in Emotion Regulation Scale (DERS) is a self-report instrument consisting of 36 items meant to measure difficulties in emotion regulation, higher scores ranging from 36- 144 indicate more significant difficulties in emotion regulation (Gratz & Roemer, 2004). We will use the cut score of 97 to identify severe difficulties in emotion regulation (Bemmouna et. Al 2022; Neacsiu et. al., 2014).
The intervention is feasible, accepted and safe - The dropout rate from treatment. | From treatment start to compleation up to 9 months.
  The dropout rate from the standard treatment, DBT- SUD skills and NET. Dropout is registered, and dichotomous variables are created (yes/no). In case of dropout, time from admission to dropout is registered.
The intervention is safe - Suicide behaviour while in treatment. | From treatment start to compleation up to 9 months.
  Prevalance of suicide behavior before treatment and while in treatment is registrert with the Columbia-suicide severity rating scale (C-SSRS) a suicidal ideation and behaviour-rating interview created to evaluate suicide risk. The interview consists of 10 categories with binary responses (yes/no) to indicate a presence or absence of the behaviour. The outcome of the C-SSRS is a numerical score obtained from the categories (Posner et.al. 2011). The participants Answer the interview 5 weeks from treatment start and at treatment compleation.
The intervention is safe - Self-harm behaviour while in treatment. | From treatment start to compleation up to 9 months.
  Prevelance of Self-harm behaviour before tratment and while in treatment is registrert with The Deliberate Self-Harm Inventory (DSHI). DSHI is a 17 -item behaviourally based, self-report instrument to assess deliberate self-harm (Gratz, 2001). In this project we create a continuous variable on frequency of self-harm behaviour and a dichotomous variable on presence of self-harm (Yes/No). e of the C-SSRS is a numerical score obtained from the categories (Posner et.al. 2011). The participants answer the DSHI at 5 weeks from treatment start and at treatment compleation.
The intervention is accepted - participation in DBT-SUD skills sessions. | From treatment start to compleation up to 9 months.
  The percentage of DBT-SUD skills sessions participated in, as well as the percentage completion of homework.
The intervention is feasible and accepted - Objective experience of treatment. | From treatment start to treatment compleation up to 9 months.
  A self-rapport questionnaire is designed to evaluate the experience of the treatment. Rating on a 5 Likert scale how different elements of the treatment are experienced on a 5-point scale. There are also open-ended questions about what in the treatment is most useful and what was the least helpful (see attachment 1-2 in protocol)

SECONDARY OUTCOMES:
The potential benefits of the intervention - Change in PTSD symptoms from base line to 3-and 12 month follow up. | From 5 weeks after admission to treatment to 12-month follow upp after treatment completion. Up to 21 months.
  Evaluate the change post-treatment and at 3 and 12 months follow up, from baseline in PTSD symptom severity, measured with PTSD Checklist for DSM-5 (PCL-5), a self-report instrument developed for quick screening of PTSD symptoms. Sum scores range from 0-80, with a score over 33 indicating the presence of PTSD (Weathers et al., 2013).
The potential benefits of the intervention - Change in Difficulties in emotion regulation from baseline to 3- to 12- month follow up. | From 5 weeks after admission to treatment to 12-month follow upp after treatment completion. Up to 21 months.
  difficulties in emotion regulation measured with Difficulties in Emotion Regulation Scale (DERS) a self-report instrument consisting of 36 items meant to measure difficulties in emotion regulation, higher scores ranging from 36- 144 indicate more significant difficulties in emotion regulation (Gratz & Roemer, 2004). We will use the cut score of 97 to identify severe difficulties in emotion regulation (Bemmouna et. Al 2022; Neacsiu et. al., 2014).
The potential benefits of the intervention - Relapse to alcohol abuse at 3- and 12-months follow up. | From treatment completion to 3- and 12 month follow up - up to 12 months.
  Alcohol Use Disorders Identification Test (AUDIT) is a 10-item screening instrument to assess severity of alcohol consumption, drinking behaviours, and alcohol-related problems. Audit scores range from 0-40 with higher scores indicating greater problems related to alcohol consumptions (Aasland, Amundsen, Bovi, Fauske & Mørland, 1990). In this project, the consumption score (question 1) with cut-of score 3 and over (drinking alcohol 2 -3 times a week) is coded into a dichotomous variable of current alcohol use (yes/no) and sum score used to assess severity of alcohol related problems. At 3 months or 12 months evaluation a cut-off score 3 and over on question 1 is registered as relapse.
The potential benefits of the intervention - Relapse to substance abuse at 3- and 12-month follow up. | From treatment completion to 3- and 12 month follow up - up to 12 months.
  Realalse to substance abuse is evaluated with the Drug Use Disorder Identification Test (DUDIT), a nine item self-report instrument developed for identification of individuals with drug-related problems. DUDIT scores range from 0-44 with higher scores indicating more drug use and drug related problems (Berman, Palmstierna, Källmén, & Bergman, 2007). In this project, the substance use frequency score (question 1) is used to identify current substance use with cut-off score score 3 and over (using substances 2-3 times a week) will be coded into a dichotomous variable (yes/no). The sum score is used to assess severity of substance related problems. At 3 months or 12 months evaluation a cut-off score 3 and over on question 1 is registered as relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Egil Jonsbu, Study Director — Norwegian University of Science and Technology; Johanna Vigfusdottir, Principal Investigator — Norwegian University of Science and Technology; Edvard Breivik, Principal Investigator — Norwegian University of Science and Technology; Erlend Mork, Study Chair — Oslo University Hospital; Lars Lien, Study Chair — National Competence Center for Co-Occurring Addictive and Psychiatric Disorders; Håkon Stenmark, Study Chair — Regional Center for Violence and Traumatic Stress and St. Olavs Hospital
Locations (1):
- Molde Treatment Center, Møre and Romsdal Hospital Trust, Molde, Møre and Romsdal, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aasland OG, Amundsen A, Bovim G, Fauske S, Morland J. [Identification of patients at risk of alcohol related damage]. Tidsskr Nor Laegeforen. 1990 May 10;110(12):1523-7. Norwegian. PMID 2339403
- [Background] Battle DE. Diagnostic and Statistical Manual of Mental Disorders (DSM). Codas. 2013;25(2):191-2. doi: 10.1590/s2317-17822013000200017. No abstract available. PMID 24413388
- [Background] Bemmouna D, Coutelle R, Weibel S, Weiner L. Feasibility, Acceptability and Preliminary Efficacy of Dialectical Behavior Therapy for Autistic Adults without Intellectual Disability: A Mixed Methods Study. J Autism Dev Disord. 2022 Oct;52(10):4337-4354. doi: 10.1007/s10803-021-05317-w. Epub 2021 Oct 9. PMID 34626285
- [Background] Berman AH, Palmstierna T, Kallmen H, Bergman H. The self-report Drug Use Disorders Identification Test: Extended (DUDIT-E): reliability, validity, and motivational index. J Subst Abuse Treat. 2007 Jun;32(4):357-69. doi: 10.1016/j.jsat.2006.10.001. Epub 2006 Dec 11. PMID 17481459
- [Background] Brady, K. T., Back, S. E., & Coffey, S. F. (2004). Substance abuse and posttraumatic stress disorder. Current directions in psychological science, 13(5), 206-209.
- [Background] Chesney E, Goodwin GM, Fazel S. Risks of all-cause and suicide mortality in mental disorders: a meta-review. World Psychiatry. 2014 Jun;13(2):153-60. doi: 10.1002/wps.20128. PMID 24890068
- [Background] Elbert, T., Hermenau, K., Hecker, T., Weierstall, R., & Schauer, M. (2012). FORNET: Behandlung von traumatisierten und nicht-traumatisierten Gewalttätern mittels Narrativer Expositionstherapie.
- [Background] Elbert, T., Schauer, M., & Neuner, F. (2015). Narrative exposure therapy (NET): Reorganizing memories of traumatic stress, fear, and violence. In Evidence based treatments for trauma-related psychological disorders (pp. 229-253). Springer, Cham.
- [Background] Espie CA, Farias Machado P, Carl JR, Kyle SD, Cape J, Siriwardena AN, Luik AI. The Sleep Condition Indicator: reference values derived from a sample of 200 000 adults. J Sleep Res. 2018 Jun;27(3):e12643. doi: 10.1111/jsr.12643. Epub 2017 Nov 29. PMID 29193493
- [Background] Goodman LA, Corcoran C, Turner K, Yuan N, Green BL. Assessing traumatic event exposure: general issues and preliminary findings for the Stressful Life Events Screening Questionnaire. J Trauma Stress. 1998 Jul;11(3):521-42. doi: 10.1023/A:1024456713321. PMID 9690191
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Gratz, K. L. (2001). Measurement of deliberate self-harm: Preliminary data on the Deliberate Self-Harm Inventory. Journal of psychopathology and behavioral assessment, 23(4), 253-263.
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of psychopathology and behavioral assessment, 26(1), 41-54.
- [Background] Grubaugh AL, Magruder KM, Waldrop AE, Elhai JD, Knapp RG, Frueh BC. Subthreshold PTSD in primary care: prevalence, psychiatric disorders, healthcare use, and functional status. J Nerv Ment Dis. 2005 Oct;193(10):658-64. doi: 10.1097/01.nmd.0000180740.02644.ab. PMID 16208161
- [Background] Harder DW, Cutler L, Rockart L. Assessment of shame and guilt and their relationships to psychopathology. J Pers Assess. 1992 Dec;59(3):584-604. doi: 10.1207/s15327752jpa5903_12. PMID 1487811
- [Background] Hogue A, Schumm JA, MacLean A, Bobek M. Couple and family therapy for substance use disorders: Evidence-based update 2010-2019. J Marital Fam Ther. 2022 Jan;48(1):178-203. doi: 10.1111/jmft.12546. Epub 2021 Aug 25. PMID 34435387
- [Background] Kopelowicz A, Ventura J, Liberman RP, Mintz J. Consistency of Brief Psychiatric Rating Scale factor structure across a broad spectrum of schizophrenia patients. Psychopathology. 2008;41(2):77-84. doi: 10.1159/000111551. Epub 2007 Nov 23. PMID 18033976
- [Background] Kroenke K. & Spitzer R.L. (2002) The PHQ-9: a new depression diagnostic and severity measure. Psychiatric Annals 32:509-521.
- [Background] Linehan, M. (2014). DBT? Skills training manual. Guilford Publications.
- [Background] Linehan, M. M. (1993). Skills training manual for treating borderline personality disorder. Guilford Press.
- [Background] Lopez-Castro T, Smith KZ, Nicholson RA, Armas A, Hien DA. Does a history of violent offending impact treatment response for comorbid PTSD and substance use disorders? A secondary analysis of a randomized controlled trial. J Subst Abuse Treat. 2019 Feb;97:47-58. doi: 10.1016/j.jsat.2018.11.009. Epub 2018 Nov 24. No abstract available. PMID 30577899
- [Background] McGovern MP, Carroll KM. Evidence-based practices for substance use disorders. Psychiatr Clin North Am. 2003 Dec;26(4):991-1010. doi: 10.1016/s0193-953x(03)00073-x. PMID 14711132
- [Background] Mills KL, Teesson M, Ross J, Peters L. Trauma, PTSD, and substance use disorders: findings from the Australian National Survey of Mental Health and Well-Being. Am J Psychiatry. 2006 Apr;163(4):652-8. doi: 10.1176/ajp.2006.163.4.652. PMID 16585440
- [Background] Najavits, L. M. (2014). Creating change: A new past-focused model for trauma and substance abuse. In P. Ouimette & J. P. Read (Eds.), Trauma and substance abuse: Causes, consequences, and treatment of comorbid disorders (2nd ed., pp. 281-303). American Psychological Association. https://doi.org/10.1037/14273-014
- [Background] Najavits LM, Schmitz M, Gotthardt S, Weiss RD. Seeking Safety plus Exposure Therapy: an outcome study on dual diagnosis men. J Psychoactive Drugs. 2005 Dec;37(4):425-35. doi: 10.1080/02791072.2005.10399816. PMID 16480170
- [Background] Post-traumatic stress disorder. London: National Institute for Health and Care Excellence (NICE); 2018 Dec. Available from http://www.ncbi.nlm.nih.gov/books/NBK542453/ PMID 31211536
- [Background] Neacsiu AD, Eberle JW, Kramer R, Wiesmann T, Linehan MM. Dialectical behavior therapy skills for transdiagnostic emotion dysregulation: a pilot randomized controlled trial. Behav Res Ther. 2014 Aug;59:40-51. doi: 10.1016/j.brat.2014.05.005. Epub 2014 May 27. PMID 24974307
- [Background] Otto MW, Hearon BA, McHugh RK, Calkins AW, Pratt E, Murray HW, Safren SA, Pollack MH. A randomized, controlled trial of the efficacy of an interoceptive exposure-based CBT for treatment-refractory outpatients with opioid dependence. J Psychoactive Drugs. 2014 Nov-Dec;46(5):402-11. doi: 10.1080/02791072.2014.960110. PMID 25364993
- [Background] Ouimette PC, Brown PJ, Najavits LM. Course and treatment of patients with both substance use and posttraumatic stress disorders. Addict Behav. 1998 Nov-Dec;23(6):785-95. doi: 10.1016/s0306-4603(98)00064-1. PMID 9801716
- [Background] Ouimette, P., Moos, R. H., & Brown, P. J. (2003). Substance use disorder-posttraumatic stress disorder comorbidity: A survey of treatments and proposed practice guidelines. In P. Ouimette & P. J. Brown (Eds.), Trauma and substance abuse: Causes, consequences, and treatment of comorbid disorders (pp. 91-110). American Psychological Association. https://doi.org/10.1037/10460-005
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Roberts NP, Roberts PA, Jones N, Bisson JI. Psychological therapies for post-traumatic stress disorder and comorbid substance use disorder. Cochrane Database Syst Rev. 2016 Apr 4;4(4):CD010204. doi: 10.1002/14651858.CD010204.pub2. PMID 27040448
- [Background] Roemer, L., Litz, B. T., Orsillo, S. M., & Wagner, A. W. (2001). A preliminary investigation of the role of strategic withholding of emotions in PTSD. Journal of Traumatic Stress, 14(1), 149-156.
- [Background] Saraiya T, Lopez-Castro T. Ashamed and Afraid: A Scoping Review of the Role of Shame in Post-Traumatic Stress Disorder (PTSD). J Clin Med. 2016 Nov 1;5(11):94. doi: 10.3390/jcm5110094. PMID 27809274
- [Background] Sinha R. Stress and addiction: a dynamic interplay of genes, environment, and drug intake. Biol Psychiatry. 2009 Jul 15;66(2):100-1. doi: 10.1016/j.biopsych.2009.05.003. No abstract available. PMID 19555787
- [Background] Stenmark H, Guzey IC, Elbert T, Holen A. Gender and offender status predicting treatment success in refugees and asylum seekers with PTSD. Eur J Psychotraumatol. 2014 Jan 30;5. doi: 10.3402/ejpt.v5.20803. eCollection 2014. PMID 24494062
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Taylor CT, Laposa JM, Alden LE. Is avoidant personality disorder more than just social avoidance? J Pers Disord. 2004 Dec;18(6):571-94. doi: 10.1521/pedi.18.6.571.54792. PMID 15615668
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Tull MT, Gratz KL, Coffey SF, Weiss NH, McDermott MJ. Examining the interactive effect of posttraumatic stress disorder, distress tolerance, and gender on residential substance use disorder treatment retention. Psychol Addict Behav. 2013 Sep;27(3):763-73. doi: 10.1037/a0029911. Epub 2012 Sep 3. PMID 22946858
- [Background] van de Glind G, van den Brink W, Koeter MW, Carpentier PJ, van Emmerik-van Oortmerssen K, Kaye S, Skutle A, Bu ET, Franck J, Konstenius M, Moggi F, Dom G, Verspreet S, Demetrovics Z, Kapitany-Foveny M, Fatseas M, Auriacombe M, Schillinger A, Seitz A, Johnson B, Faraone SV, Ramos-Quiroga JA, Casas M, Allsop S, Carruthers S, Barta C, Schoevers RA; IASP Research Group; Levin FR. Validity of the Adult ADHD Self-Report Scale (ASRS) as a screener for adult ADHD in treatment seeking substance use disorder patients. Drug Alcohol Depend. 2013 Oct 1;132(3):587-96. doi: 10.1016/j.drugalcdep.2013.04.010. Epub 2013 May 6. PMID 23660242
- [Background] Van IJzendoorn, M. H., & Schuengel, C. (1996). The measurement of dissociation in normal and clinical populations: Meta-analytic validation of the Dissociative Experiences Scale (DES). Clinical Psychology Review, 16(5), 365-382.
- [Background] Vanderplasschen W, Vandevelde S, Broekaert E., (2014). Therapeutic communities for treating addictions in Europe. Evidence, current practices and future challenges. Luxembourg: Publications Office of the European Union.
- [Background] Vigfusdottir, J., Hoidal, R., Breivik, E., Jonsbu, E., Dale, K. Y. & Mork, E. (2023). The Norwegian version of the Personal Feelings Questionnaire-2: The translation, clinical utility, and psychometric properties. Manuscript submitted for publication.
- [Background] Vigfusdottir, J., Dale, K. Y., Gratz, K. L., Klonsky, E. D., Jonsbu, E., & Høidal, R. (2020). The psychometric properties and clinical utility of the Norwegian versions of the deliberate self-harm inventory and the inventory of statements about self-injury. Current Psychology, 1-11.
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] Weathers, F. W., Litz, B. T., Keane, T. M., Palmieri, P. A., Marx, B. P., & Schnurr, P. P. (2013). The ptsd checklist for dsm-5 (pcl-5). Scale available from the National Center for PTSD at www. ptsd. va. gov, 10.
- [Background] Westphal, M., Aldao, A., & Jackson, C. (2017). Emotion dysregulation in comorbid posttraumatic stress disorder and substance use disorders: A narrative review. Military Psychology, 29(3), 216-233.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT06345053/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT06345053/ICF_001.pdf